CLINICAL TRIAL: NCT04993963
Title: Impact of Prehabilitation on the Quality of Recovery (QoR) After Heart Valve Surgery.
Brief Title: Prehabilitation and Heart Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rec/00881 Tayyaba kiran
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Valvular Heart Disease
Keywords: prehabilitation; quality of recovery; heart valve surgery
MeSH Terms: conditions — Heart Valve Diseases | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycle Ergometery Training (Prehabilitation) (Experimental): Hospital-based ergometer cycling for 20 minutes (Including warm-up and cooldown) Interval training on cycle ergometer: between 40% and 60% Vo2max, perceived exertion <13 on Borg scale
  Interventions: Other: Cycle Ergometery Training (Prehabilitation)
- Control Standard Group (Active Comparator): Breathing exercise 15 Reps and Walk (10-15 minutes)
  Interventions: Other: Control Standard Group

INTERVENTIONS:
Other: Cycle Ergometery Training (Prehabilitation) — Interval training on cycle ergometer: between 40% and 60% Vo2max, perceived exertion <13 on Borg scale 20-30 min/session/day (intermittent of exercise 2-3 mint, followed by 1-2 min of active recovery) Cool down (5 minutes) AROM +Body stretch
  Arms: Cycle Ergometery Training (Prehabilitation)
Other: Control Standard Group — Breathing exercise 15 Reps and Walk (10-15 minutes)
  Arms: Control Standard Group

SUMMARY:
To evaluate the impact of prehabilitation on quality of recovery in heart valve surgery. To evaluate the effects of Mild to moderate valvular diseases with Newyork Heart Association (NYHA) grade I and II . Previous studies were designed to target on Coronary artery bypass graft surgery (CABGs) patients no specifically heart valve surgery patients was studied so this study cover this aspect as well so from the outcomes of this study we will determine the prehabilitation effects on valvular surgery patients.

DETAILED DESCRIPTION:
A review stated that " the concept of prehabilitation has entered the forefront which encompasses multidisciplinary interventions to improve health and lessen the incidence of postoperative decline.

In the previous study held in pre-operative assessment clinic between March 2016 and August 2016, evaluated that PREHAB programme for frail patients undergoing CABG or Valve surgery may be able to improve functional ability and reduce hospital length of stay for those patients undergoing cardiac surgery.

previous other studies, parental study which is PREQUEL study recruitment started in July 2018 expect patient recruitment and 3 months of follow-up will be completed in June 2022 then their analysis will be done.

To improve functional and enhance the resources and postoperative recovery, prehabilitation plays a very cardial role. In some studies, it has been noticed that preoperative improvement in physical fitness, improve functional capacity all this is the part of the model for improving post-surgery recovery, this could play a vital role.

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting heart valve surgery for repair or replacement
* Both gender
* Mild to moderate valvular diseases
* NYHA grade I and II
* Pre-frail to moderately frail patients with a CFS of 4-6
* Patients with an estimated 6-8 weeks of surgical waiting list time.
* Able to perform 6MWT at baseline with RPE<13

Exclusion Criteria:

* Patients with severe left ventricular obstructive disease (severe aortic or mitral stenosis and dynamic left ventricular outflow obstruction).
* Patients with unstable or recently unstable cardiac syndrome
* Other than valve surgeries e.g. CABG
* Hospitalization for arrhythmias/ congestive heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | After 6 weeks, 1 month after CABG
  15-item Quality of Recovery (QoR-15) is one of the standardized outcomes for assessing patient comfort after surgery. The QoR-15 score includes the items measuring pain, physical comfort, physical independence, psychological support, and emotional state. The QoR-15 score runs from 0 to 150. Higher scores indicate better Quality of life.
Clinical Frailty Score | After 6 weeks, 1 month after CABG
  Frailty is a valid and clinically important construct that is recognizable by physicians. Clinical judgments about frailty can yield useful predictive information. Initial Clinical Frailty Scale assessment had access to diagnoses and assessments related to these variables and other measures of comorbidity, function, and associated features that inform clinical judgments about the severity of frailty. It was modified to a 9-point scale to include very severely frail and terminally ill. It evaluates specific domains, including comorbidity, function, and cognition, to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Pakistan Institute of medical sciences (PIMS), Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milder DA, Pillinger NL, Kam PCA. The role of prehabilitation in frail surgical patients: A systematic review. Acta Anaesthesiol Scand. 2018 Nov;62(10):1356-1366. doi: 10.1111/aas.13239. Epub 2018 Aug 10. PMID 30094821
- [Background] McCann M, Stamp N, Ngui A, Litton E. Cardiac Prehabilitation. J Cardiothorac Vasc Anesth. 2019 Aug;33(8):2255-2265. doi: 10.1053/j.jvca.2019.01.023. Epub 2019 Jan 12. PMID 30765210
- [Background] Steinmetz C, Bjarnason-Wehrens B, Baumgarten H, Walther T, Mengden T, Walther C. Prehabilitation in patients awaiting elective coronary artery bypass graft surgery - effects on functional capacity and quality of life: a randomized controlled trial. Clin Rehabil. 2020 Oct;34(10):1256-1267. doi: 10.1177/0269215520933950. Epub 2020 Jun 16. PMID 32546065
- [Background] Norris CM, Close JCT. Prehabilitation for the Frailty Syndrome: Improving Outcomes for Our Most Vulnerable Patients. Anesth Analg. 2020 Jun;130(6):1524-1533. doi: 10.1213/ANE.0000000000004785. PMID 32384342